CLINICAL TRIAL: NCT05429281
Title: Comparative Efficacy of Pilates-Based Core Strengthening, Plyometric-Based Muscle Loading, and Their Combination on Postural Control, Balance, and Mobility in Children With Unilateral Cerebral Palsy
Brief Title: The Role of Pilates, Plyometrics, and Their Combination for Children With Unilateral Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0021/0114
Record Dates: First submitted 2022-06-18; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: A prospective, assessor-blinded, randomized study
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blinded to the treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pilates-based Core Strengthening Group (Active Comparator): Participants in this group performed eight PsCS exercises geared predominantly to the core muscles.
  Interventions: Other: Pilates-based Core Strengthening Exercises
- Plyometric-based Muscle Loading Group (Active Comparator): Participants in this group performed 10 PlyoML exercises primarily focused on the lower body.
  Interventions: Other: Plyometric-based Muscle Loading Exercises
- Combined training group (Experimental): Participants in this group performed the same exercises as the PsCS and PlyoML groups, although with half the number of sets/repetitions.
  Interventions: Other: Combined Pilates and Plyometrics

INTERVENTIONS:
Other: Pilates-based Core Strengthening Exercises — The PsCS group performed eight Pilates exercises over 45 minutes, three times per week for 12 successive weeks. The training was conducted under the supervision of a physical therapist who had more than 5 years of experience in Pilates.
  Arms: Pilates-based Core Strengthening Group
Other: Plyometric-based Muscle Loading Exercises — The PlyoML group performed 10 plyometric exercises over 45 minutes, three times per week for 12 successive weeks. The training was conducted under the close supervision of a licensed pediatric physical therapist. The safety and performance guidelines, defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association, were considered during training.
  Arms: Plyometric-based Muscle Loading Group
Other: Combined Pilates and Plyometrics — The combined training group performed the same exercises as the PsCS and PlyoML groups, although with half the number of sets/repetitions over 45 minutes, three times per week for 12 successive weeks. The PsCS and PlyoML were executed within the same session, with a 10-to-15-minute rest interval. The training was conducted under the close supervision of a licensed pediatric physical therapist. The safety and performance guidelines, defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association, were considered during training.
  Arms: Combined training group

SUMMARY:
This study was conducted to compare the effect of Pilates-based core strengthening (PsCS) and plyometric-based muscle loading (PlyoML) and their combination on postural control, balance, and mobility in children with unilateral cerebral palsy (ULCP). Eighty-one children with ULCP were randomly allocated to the PsCS (n = 27), PlyoML (n = 27), or combined intervention (n = 27) group. Participants in the three groups were assessed for postural control, balance, and mobility on the pre and post-treatment occasions.

DETAILED DESCRIPTION:
Eighty-one children with ULCP were recruited from the Physical Therapy Outpatient Clinic of College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, King Khalid Hospital, and a tertiary referral hospital, Al-Kharj, Saudi Arabia. Their age ranged between 12 and 18 years, were functioning at levels I or II according to the Gross Motor Function Classification System, and had spasticity levels 1 or 1+ per the Modified Ashworth Scale. Children were excluded if they had fixed deformities, underwent neuromuscular or orthopedic surgery in the last 12 months, submitted to BOTOX injection in the past 6 months, had attentional neglect, and if they had cardiopulmonary problems preventing them from performing high-intense exercise training.

Outcome measures

* Postural control: The directional dynamic limit of stability (forward, backward, paretic, and non-paretic) and overall limit of stability were assessed using the Biodex balance system.
* Balance and mobility: The Community Balance and Mobility Scale (CB&M), Functional Walking Test (FWT), and Timed Up and Down Stair test (TUDS) were used to quantify balance and mobility capacity.

Interventions

All groups were trained for 45 minutes, twice per week, for 12 successive weeks. The PsCS group performed eight Pilates exercises geared predominantly toward the core muscles. The PlyoML group performed 10 plyometric exercises primarily focused predominantly on the lower body. The combined group combined the same exercises as the PsCS and PlyoML groups, although with half the number of sets/repetitions.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral cerebral palsy
* Age 12-18 years
* Motor function level I or II according to the Gross Motor Function Classification System.
* Spasticity level 1 or 1+ according to the Modified Ashworth Scale

Exclusion Criteria:

* Structural deformities/contractures
* Musculoskeletal or neural surgery in the last year
* BOTOX injection in the last 6 months.
* Cardiopulmonary disorders interfere with the ability to engage in exercise training.
* Perceptual and/or behavioral disorders.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 81 (Actual)
Dates: Start 2021-02-07 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Limit of postural stability | 2 months
  The capacity to control and move the center of gravity in various directions across their base of support was assessed utilizing the Biodex balance system. Values are expressed as accuracy % and higher scores mean better balance capability.

SECONDARY OUTCOMES:
Community Balance and Mobility Scale | 2 months
  Community Balance and Mobility Scale is a performance-based measure assessing high-level balance capabilities while also addressing the speed and coordination components necessary for the ordinary community function.
  The scale consists of 13 items. Item scores range from zero (complete inability of task execution) to five (the most successful task completion), and the maximum possible score is 96. A higher score indicates better performance.
Functional Walking Test | 2 months
  The Functional Walking Test is a valid and reliable measure for assessing functional waking capacity in ambulant children with cerebral palsy. The test consists of 11 items including kneel walking, transitions to standing, incline walking, ascending/descending stairs, and walking a narrow beam, all of which focus on the postural control and balance components of walking. The maximum score is 23 and higher scores indicate better walking capacity
Timed Up and Down Stair test | 2 months
  The Timed Up and Down Stairs test measures the time (in seconds) that the children take to go up a 14-step stair flight (each step was 20 cm in height), turn around, and come back down. Shorter time indicates better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia